CLINICAL TRIAL: NCT02223780
Title: Can Early Introduction of Specialized Palliative Care Limit Intensive Care, Emergency and Hospital Admissions in Patients With Severe and Very Severe COPD? A Randomized Study
Brief Title: Early Palliative Care for Patients With Severe and Very Severe COPD: a Randomised Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Jean-Paul Janssens, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Projet 13-102; 406740_145086/1 (Other Grant/Funding Number: SNF406740_145086/1)
Record Dates: First submitted 2014-08-08; First posted 2014-08-22 (Estimated); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: COPD
Keywords: COPD; palliative care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Placebo Comparator): standard management
  Interventions: Other: early palliative care
- early palliative care (Active Comparator): early palliative care
  Interventions: Other: early palliative care

INTERVENTIONS:
Other: early palliative care — the patients will benefit from an early palliative care consultation

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common and, despite existing treatment options, progressive lung disease. Patients with COPD often have only limited access to palliative care. The goal of this research project is to improve the quality of life of patients with COPD.

Background In many cases, the symptoms of advanced COPD (including shortness of breath, pain and depression) are insufficiently alleviated. In addition, often in connection with an infection, patients frequently suffer from respiratory decompensation; this may lead to invasive interventions as well as the admission to the emergency room or an intensive care unit. It may ultimately lead to the death of the patient.

Aim This study aims to show that early palliative care can reduce the number of necessary invasive interventions and improve the quality of life of patients with COPD. For this purpose, a group of patients receiving early, standardized palliative care will be compared to a group of patients receiving customary treatment only, without systematic intervention by palliative care experts.

Significance The results of this study should make it possible to efficiently use the medical resources which are required for the appropriate care of patients with COPD. The goal is the best possible quality of life and better coordination of the measures taken, especially with regard to the area of acute care and the wishes of the patient.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the effectiveness of the introduction of early specialized palliative care on hospital, intensive care unit and emergency admissions of patients with severe and very severe COPD

Secondary objectives are:

The impact of early palliative care on the mood and anxiety of patients with severe and very severe COPD The impact of early palliative care on the health-related quality of life of patients with severe and very severe COPD.

The impact of early palliative care on the prescription of antibiotics during the last month of life of patients 4. The impact of early palliative care on advance care planning and end-of-life decision-making will be compared between the two groups Methodology Randomized study to one of the two groups in a ratio without stratification.

Study Duration 3 years Study Center(s) Single-center study Number of Subjects 180 patients Intervention Early specialized palliative care intervention Significance Given the trends toward aggressive and costly care near end-of-life among patients with COPD, a timely introduction of palliative care may limit unnecessary and burdensome personal and societal costs, and invasive approaches. The results of this study may provide some direction for future palliative care interventions in this particular population

ELIGIBILITY:
Inclusion Criteria:

* COPD defined according to GOLD criteria (FEV1/FVC < 70%) stage III or IV (FEV1 < 50% predicted)

  * and/or long term treatment with either domiciliary oxygen or home mechanical ventilation
  * and or one or more hospital admissions in the previous year for an acute exacerbation

Exclusion Criteria:

* Moderate or severe cognitive impairment (MMSE<20)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
length of stay hospital, intensive care unit and emergency admissions | 1 year
  number of days

SECONDARY OUTCOMES:
depression and anxiety | 1 year
  HADS
Health related quality of life assessed by a generic questionnaire | 1 year
  SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Janssens, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Weber C, Stirnemann J, Herrmann FR, Pautex S, Janssens JP. Can early introduction of specialized palliative care limit intensive care, emergency and hospital admissions in patients with severe and very severe COPD? a randomized study. BMC Palliat Care. 2014 Oct 21;13:47. doi: 10.1186/1472-684X-13-47. PMID 25927907
- See also: link of the national fund — http://www.nfp67.ch/